CLINICAL TRIAL: NCT05597605
Title: The SHINE Study: An Open Label, Interventional, Multicentre, Prospective Feasibility Study, Designed to Evaluate the Safety of Implant and Preliminary Performance of the SHINE SYSTEM in Diabetic Subjects
Brief Title: The SHINE Study: Safety of Implant and Preliminary Performance of the SHINE SYSTEM in Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indigo Diabetes NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IND008
Record Dates: First submitted 2022-09-19; First posted 2022-10-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Ketoacidosis, Diabetic; Hyperglycaemia (Diabetic); Hypoglycemia
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Ketoacidosis; Hyperglycemia; Hypoglycemia; GCM
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Ketoacidosis; Hyperglycemia; Hypoglycemia; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The SHINE SYSTEM (Experimental)
  Interventions: Device: The SHINE SYSTEM

INTERVENTIONS:
Device: The SHINE SYSTEM — The FUSHO sensor, which is part of the SHINE SYSTEM, is a continuous multi-metabolite monitoring (CMM) sensor which is a miniaturized near-infrared spectrometer that measures the absorption of light in the interstitial fluid to quantify the concentration of multiple metabolites

SUMMARY:
The objectives of SHINE study are to confirm the safety aspects of the SHINE SYSTEM. Moreover, the goal of this clinical investigation is the initial evaluation of sensor's performance by assessing sensor's ability to qualitatively detect the appropriate analytes in subjects with diabetes of 18 years and older.

DETAILED DESCRIPTION:
Indigo Diabetes N.V. is currently developing an active implantable medical device, intended to be used for real time, continuous measurement of glucose and ketone levels in the interstitial fluid in adults (18 years and older) with diabetes mellitus. Based on the outcome of the GLOW Study, Indigo developed a prototype, the SHINE SYSTEM, that will be used during the planned clinical investigation (SHINE study).The objectives of SHINE study are to confirm the safety aspects of the SHINE system. Moreover, the goal of this clinical investigation is the initial evaluation of sensor's performance by assessing sensor's ability to qualitatively detect the appropriate analytes in subjects with diabetes of 18 years and older. Clinical performance of the device will not be formally evaluated during this clinical investigation. The study is designed to enable data collection (i.e., continuous collection of data by FUSHO sensor, implanted in study subject, combined with simultaneous collection of data collected by Dexcom G6), which will be used to develop the software algorithm in a future version of the device, in order to display measurements in real-time to the user.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to sign an informed consent form (ICF)
* Adult subjects, age ≥ 18
* Subjects willing to comply to study protocol requirements (study visits with frequent venous blood sampling and deliberate insulin, glucose, ketone and lactate (sub study only) challenges)
* Subjects willing to wear a Dexcom G6 CGM during duration of the study
* Subjects willing to charge the FUSHO SENSOR/ED and CHARGER on daily basis
* Patients with type 1 diabetes mellitus (T1DM) according to WHO criteria, diagnosed for at least 12 months prior to screening, on Multiple Daily Injections (MDI), not on insulin pump treatment during the course of the study
* Patients with type 2 diabetes mellitus (T2DM) on Intensive Insulin Therapy (IIT), with a minimum of four injections per day and known dosing parameters

Exclusion Criteria:

* Known allergy to PDMS
* Subjects with a contraindication to undergo challenging tests (i.e., ischemic heart disease, epilepsy, panhypopituitarism, hypoadrenalism, untreated hypothyroidism)
* History of severe hypoglycaemia in the previous 6 months. Severe hypoglycaemia is defined as hypoglycaemia resulting in loss of consciousness or seizure
* History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months
* History of, hepatitis C or HIV or other disease transmissible by blood
* A condition requiring or likely to require magnetic resonance imaging (MRI) during the study duration
* Female subjects who are pregnant, planning on becoming pregnant or nursing
* Coagulation disorder, wound healing and bleeding disorder or taking anticoagulant medication (oral anticoagulants; antiplatelets (such as aspirin, ticagrelor are allowed).
* Anemia identified by a haemoglobin <14 g/dL for men or <12 g/dL for women
* The presence of any other active implanted device
* The presence of any other CGM sensor or transmitter located in lower abdomen or back (other location is acceptable)
* Waist circumference of >120 cm
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Primary Safety Objectives: Confirm safe implantation of the SENSOR in human subcutaneous tissue (insertion procedural safety) | 30 days
  Incidence of FUSHO SENSOR insertion procedure-related serious adverse events within 30 days from implant
Primary Safety Objectives: Confirm the safety of the device during the implantation period (safety of device integration in the subcutaneous tissue) | 6 months
  Assessment of device related adverse events during 6 months of implant use
Primary Initial Performance Objectives: Demonstration of SENSOR stability | 6 months
  Demonstrate that device is able to provide a stable spectral signal and whether it is feasible to use these data points to create an algorithm. SENSOR Stability is defined by maintaining its spectral characteristics (availability, intensity and range) over its implantation duration of 6 months
Primary Initial Performance Objectives: Confirm the ability to (a) retrieve spectral and metadata from the SENSOR and upload to the CLOUD | 6 months
  (a) Evaluation of the Bluetooth transmission: successful transmission of the spectral data from FUSHO SENSOR to the CLOUD via Bluetooth Low Energy (BLE). The proportion of data transmitted to the CLOUD versus the expected amount of data when device used as intended
Primary Initial Performance Objectives: Confirm the ability to (b) show the battery and SENSOR-ED connectivity status to subject | 6 months
  (b) Display of battery and FUSHO SENSOR-ED connectivity status to subject
Primary Initial Performance Objectives: Confirm the ability to (c) recharge the SENSOR, ED and CHARGER. | 6 months
  (c) Charging (charging efficiency) of the FUSHO SENSOR, as recorded on the APP

SECONDARY OUTCOMES:
Secondary Safety Objectives: Confirm safe explantation of the SENSOR from human subcutaneous tissue (removal procedural safety) | 30 days
  Incidence of FUSHO SENSOR removal-related serious adverse events within 30 days from explant
Secondary Safety Objectives: Confirm general safety in the clinic and during home use (general safety) | 6 months
  * All Serious Adverse Events collected throughout the study and reported at 30 days, 3 months and 6 months
  * Assessment of device related adverse events at 30 days, 3 and 6 months
  * Wound status at each visit. Final result on healing just at explant.
Secondary Performance Objective: Assessment of procedural success for the implantation procedure | 30 days
  Successful FUSHO implantation (first implant in case of re-implant) procedure on average performed within 20 minutes (from incision to closure) without occurrence of procedure related SAEs
Secondary Performance Objective: Assessment of procedural success for the explantation procedure | 30 days
  Successful FUSHO explantation procedure on average performed within 20 minutes (from incision to closure) without occurrence of procedure related SAEs
Secondary Performance Objective: Assessment of procedural success for the implantation and explantation procedure | 30 days
  Procedural success defined as implantation of the FUSHO SENSOR within an average of 20 minutes (from start incision to closing of skin) without the occurrence of procedure related adverse events up to 30 days after implant
Secondary Performance Objective: Assessment of procedural success for the implantation and explantation procedure | 30 days
  The primary initial performance endpoint at further timepoints through 30 days and 3 months

OTHER OUTCOMES:
Exploratory Analysis: Establishment of a model for evaluation of blood glucose, ketone and lactate values by the SENSOR by using the values obtained by other than SENSOR data | 6 months
  Development and refinement of a model that allows correct analysis of the spectral data read and translation into glucose, ketone and lactate (for sub-study only) values. The values will be analysed in conjunction with values obtained by comperative methods and used to further adjust this model. The model is expected to be able to demonstrate increased performance by subsequent iterations based on known absolute values. Iterations are expected to be performed until values are suitable for validation
Exploratory Analysis: Accuracy of measurements for glucose demonstrated by Mean Absolute Relative Difference (MARD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Relative Difference (MARD) intended for evaluation of the appropriateness of the algorithm/model for prediction of glucose. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for ketones demonstrated by Mean Absolute Relative Difference (MARD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Relative Difference (MARD) intended for evaluation of the appropriateness of the algorithm/model for prediction of ketones. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for lactate demonstrated by Mean Absolute Relative Difference (MARD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Relative Difference (MARD) intended for evaluation of the appropriateness of the algorithm/model for prediction of lactate. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for glucose demonstrated by Mean Absolute Deviation (MAD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Deviation (MAD) intended for evaluation of the appropriateness of the algorithm/model for prediction of glucose. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for ketones demonstrated by Mean Absolute Deviation (MAD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Deviation (MAD) intended for evaluation of the appropriateness of the algorithm/model for prediction of ketones. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for lactate demonstrated by Mean Absolute Deviation (MAD) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Mean Absolute Deviation (MAD) intended for evaluation of the appropriateness of the algorithm/model for prediction of lactate. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for glucose demonstrated by Error Grid Analysis (EGA) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Error Grid Analysis (EGA) intended for evaluation of the appropriateness of the algorithm/model for prediction of glucose. No health outcomes (e.g. ability to predict glycaemic values) are evaluated.
Exploratory Analysis: Accuracy of measurements for ketones demonstrated by Error Grid Analysis (EGA) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Error Grid Analysis (EGA) intended for evaluation of the appropriateness of the algorithm/model for prediction of ketones. No health outcomes (e.g. ability to predict glycaemic values) are evaluated
Exploratory Analysis: Accuracy of measurements for lactate demonstrated by Error Grid Analysis (EGA) | 6 months
  Post hoc analysis of accuracy of measurements for glucose demonstrated by Error Grid Analysis (EGA) intended for evaluation of the appropriateness of the algorithm/model for prediction of lactate. No health outcomes (e.g. ability to predict glycaemic values) are evaluated
Exploratory Analysis: Histopathology analysis of the biopsy | 6 months
  Histopathology analysis of the biopsy at explant on macroscopic and microscopic level, with Haematoxylin-Eosin (HE) staining, to assess potential changes of surrounding cells and tissue around the sensor and local tissue tolerance/interaction by investigating local tissue inflammation (fibrosis, foreign body reaction (e.g. presence of giant cells, macrophages and other))

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, Prof. Dr., Principal Investigator — University Hospital, Antwerp
Locations (3):
- University Hospital Àntwerp, Antwerp, Belgium
- Lapeyronie Montpellier University Hospital, Montpellier, France
- University Medical Centre, Ljubljana, Slovenia